CLINICAL TRIAL: NCT07350447
Title: Predictors of Laparoscopy Conversion in the Treatment of Adhesive Small Bowel Obstruction
Brief Title: Predictors of Laparoscopy Conversion in Adhesive Small Bowel Obstruction
Status: Not yet recruiting | Type: Observational
Sponsor: Almazov National Medical Research Centre (Other)
Responsible Party: Principal Investigator, Kotkov Pavel, Assistant professor of the general surgery department, Almazov National Medical Research Centre
Other Study IDs: 14071979
Record Dates: First submitted 2025-12-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: Adhesive small bowel obstruction; Ahesiolysis; Laparoscopic adhesiolysis; abdominal adhesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopy group: Patients with acute adhesive intestinal obstruction, operated through surgical intervention, that was initiated and completed using endovideosurgical methods.
  Interventions: Procedure: Laparoscopic adhesiolysis
- Conversion group: Patients with acute adhesive intestinal obstruction, in whom surgical intervention was initiated by endovideosurgical means, however, during the operation there was a need for laparotomy and the surgical procedure was completed by laparotomy access.
  Interventions: Procedure: Laparotomic adhesiolysis

INTERVENTIONS:
Procedure: Laparoscopic adhesiolysis — Dissection of intra-abdominal adhesions performed laparoscopically in accordance with the principles adopted in the medical institution.
  Groups: Laparoscopy group
Procedure: Laparotomic adhesiolysis — Traditional adhesiolysis, performed via laparotomy after unsuccessfull attempt of endovideosurgical approach.
  Groups: Conversion group

SUMMARY:
The goal of this observational study is to reveal predictors of unsuccessfull laparoscopic intervention in adult patients with adhesive small bowel obstruction. The main question it aims to answer is: are there any strong predictors of laparoscopy conversion in patients with small bowel obstruction, caused by intraabdominal adhesions.

DETAILED DESCRIPTION:
Considering the undeniable advantages of laparoscopic interventions over laparotomic ones, the question of choosing a surgical approach in patients with acute adhesive intestinal obstruction can be reformulated as follows: in what situations is endovideosurgical intervention generally appropriate and feasible? A laparoscopic approach to severely distended bowel loops and widespread adhesions may increase the risk of serious complications. Indeed, some authors report intestinal injury in 6.3-26.9% of patients undergoing laparoscopic adhesiolysis for acute adhesive intestinal obstruction, which is statistically significantly higher than the same rate in patients operated on using a traditional approach. Therefore, a priority should be addressing the issue of adequately selecting patients who, based on a number of clinical indicators, are suitable for laparoscopic surgery or, at least, have no contraindications. While some parameters, such as acute cardiovascular or respiratory failure and pregnancy in the third trimester, can be defined as absolute contraindications to endovideosurgical access, a number of clinical and instrumental indicators are debatable. Despite the fact that this issue has been extensively covered in the literature, and the list of predictors of unsuccessful laparoscopic adhesiolysis is currently quite impressive, a standardized approach to access selection is lacking or is determined largely intuitively.

The aim of this work is to determine reliable anamnestic, clinical and instrumental signs that would indicate a high risk of conversion of the laparoscopic intervention in patients with acute adhesive intestinal obstruction.

The study is planned to be a multicenter, retrospective case-control study. Clinical data will be collected at four medical institutions in St. Petersburg. The medical records of patients who underwent emergency and urgent surgery for acute adhesive intestinal obstruction will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent emergency and urgent surgery for acute adhesive intestinal obstruction
* the surgery was performed laparoscopically
* the surgery was initiated laparoscopically and completed via laparotomy

Exclusion Criteria:

* acute adhesive intestinal obstruction in the hernial sac
* pregnant in the third trimester
* patients with severe cardiovascular or respiratory failure
* patients with hemodynamic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, operated in surgical departments of 4 different hospitals in Saint-Petersburg and one hospital in Perm, Kazan and Yekaterinburg respectively.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of succesfull laparoscopic interventions | At the discharge from the hospital (assessed up to 10 days)
  The ratio of successful laparoscopic interventions to the total number of operations

SECONDARY OUTCOMES:
Diameter of intestinal loops | Perioperative
  Diameter of intestinal loops (cm), ascertained during X-ray treatment before the operation. The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Known or suspected complex adhesive process | Perioperative
  Presence of known or suspected complex adhesive process (according to anamnestic data). The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Number of laparotomy operations | Perioperative
  Number of laparotomy operations according to anamnestic data. The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Ischemia or necrosis of the intestine | Perioperative
  Ischemia or necrosis of the intestine, requiring resection (diagnosed intraoperatively). The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Obstruction level | Perioperative
  Obstruction level measured in cm from Treitz ligament to obstruction site, diagnosed intraoperatively. The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Duration of acute intestinal obstruction | Perioperative
  Duration of acute intestinal obstruction, measured in hours from pain onset till surgery. The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.
Time of day at the start of the surgical intervention | Perioperative
  Time of day at the start of the surgical intervention, specified as daytime (from 9:00 to 18:00), evening (from 18:00 to 24:00), night (from 24:00 to 9:00). The correlation between this outcome and the likelihood of unsuccessful laparoscopic adhesiolysis and the need for laparotomy will be studied. The power of corellation will be measured according to the Spearman correlation coefficient and relative risk with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel А Kotkov, MD, Principal Investigator — Almazov National Medical Research Centre
Locations (7):
- Russia (7):
  - Kazan Federal University, Kazan'
  - City Clinical Hospital No. 4, Perm
  - Almazov National Medical Research Centre, Saint Petersburg
  - Mariinskaya Hospital, Saint Petersburg
  - Saint-Petersburg I.I. Dzhanelidze research institute of emergency medicine, Saint Petersburg
  - The City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - City Clinical Hospital No. 40, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Undecided